CLINICAL TRIAL: NCT03666598
Title: The Effects of a Tourniquet on Implant Migration and Muscle Strength and Function in Patients Operated With Total Knee Arthroplasty
Brief Title: The Effects of a Tourniquet in Total Knee Arthroplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Zimmer Biomet (Industry); University of British Columbia (Other); Karolinska University Hospital (Other); St. Olavs Hospital (Other); Kristiansund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/2206
Record Dates: First submitted 2018-08-30; First posted 2018-09-12 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasty, Replacement, Knee; Tourniquets; Pain, postoperative; Muscle strength
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No tourniquet (No Intervention): No use of tourniquet during surgery
- Tourniquet (Experimental): Use of tourniquet during surgery. The cuff will be inflated to 300mmHg
  Interventions: Device: Tourniquet

INTERVENTIONS:
Device: Tourniquet — In the patients randomized to the use of tourniquet, the tourniquet time starts before skin incision and terminates when the wound closure starts. The cuff pressure is set at 300mmHg.
  Arms: Tourniquet

SUMMARY:
About 5000 total knee arthroplasties (TKA) are performed annually in Norway. Pain and reduced physical function is present in patients operated with TKA up to a year after surgery and about one of five patients are not satisfied with the outcome from TKA surgery. The use of tourniquet during surgery may also have impact on pain and physical function. Whether TKA surgery should be performed with or without the use of tourniquet, is a much-debated issue in orthopedic surgery today, and there is still no consensus in this field. This study will investigate early muscle strength and power recovery, neuromuscular recordings, neuronal changes and patient reported outcome measures after surgery with tourniquet versus not tourniquet.The findings in this study are expected to have implications for rehabilitation and the outcome of the TKA surgery.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthrosis qualifying for total knee arthroplasty

Exclusion Criteria:

* Coagulation disease
* Rheumatoid arthritis
* Peripheral vascular disease
* Malign disease
* Pregnancy
* On-going infection
* Not able to understand written and oral information in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mmax | Change from 1) preoperative (baseline) to day 2 postoperative, 2) change from preoperative to 8 weeks postoperative, 3) change from preoperative to 1 year postoperative
  EMG recordings are made using 10mm electrodes (Ag-AgCl) attached in a bipolar configuration over the vastus lateralis and rectus femoris
Nerve growth factor (NGF) | Change from during surgery to 8 weeks postoperative
  Analysis from muscle biopsies harvested from the m. vastus lateralis
Forgotten Joint Score | Change from 1) preoperative (baseline) to 2) change from preoperative to 8 weeks postoperative, 3) change from preoperative to 1 year postoperative
  The stair climbing test measures the time (in seconds) to ascend, turn around and descend a regular stairway of 11 steps. The patients are asked to perform the test as quickly as possible.

SECONDARY OUTCOMES:
Maximal leg strength | Change from 1) preoperative (baseline) to day 2 postoperative, 2) change from preoperative to 8 weeks postoperative, 3) change from preoperative to 1 year postoperative
  1RM leg strength is measured using a leg press ergometer with the participant in a supine position (Steens Physical; Ring Mekanikk, Moelv, Norway)
Maximal knee extension strength | Change from 1) preoperative (baseline) to day 2 postoperative, 2) change from preoperative to 8 weeks postoperative, 3) change from preoperative to 1 year postoperative
  1RM knee extension is measured using a knee extension equipment (Body-Solid, Forest Park, IL, USA) with the participant in a seated position.
Rate of force development, voluntary activation and muscle contractility | Change from 1) preoperative (baseline) to day 2 postoperative, 2) change from preoperative to 8 weeks postoperative, 3) change from preoperative to 1 year postoperative
Daily physical activity | Change from day 3 - 10 postoperative to 1 year postoperative (1 week measurement)
  Body worn activity monitor
EuroQual 5D-L | Preoperative, 8 weeks, 1 year postoperative
  Patient reported outcome measure
Numeric Rating Scale (NRS) | Preoperative, from day 1 postoperative to 4 weeks postoperative, 8 weeks and 1 years postoperative
  Evaluating pain. The scale range from 0 (no pain) to 10 (worst pain imaginable) (7). The patients are asked to write down NRS values both at rest and during activity each day for the first 4 weeks postoperatively in a home log.
Hemoglobin values | Preoperatively, day 1 postoperative
  g/dL
Volume of bleeding | During surgery and day 1 postoperative
  Total volume of bleeding during surgery and in the drain
Length of hospital stay | From day of surgery until 10 days postoperative
  Number of days
Knee circumference | Preoperative and day 1 postoperative
  The circumference of the knee is measured 1 cm proximal to the patella base
Knee joint range of motion | Preoperative, 1 day, 8 weeks,1 year postoperative
  Maximal flexion and extension
Forgotten Joint Score | Preoperative, 8 weeks, 1 year postoperative
  Patient reported outcome measure
Gene expression analyses. RT-PCR for expression levels for VEGF, NGF, SP, CGRP, IL-6, IL-1, TNF-alpha, Bad, Bax, Bid, Bim, Fas, Fas-ligand, Bcl-2, Mcl, and FLIP. Results will be normalized to GAPDH expression levels. | Peroperative and 8 weeks postoperative
  Analysis from muscle biopsies harvested from the vastus lateralis (muscle)
Neuronal markers; PGP, GAP-43 | During surgery and 8 weeks postoperative
  Analysis from muscle biopsies harvested from the vastus lateralis (muscle)
Neuromediators; SP, CGRP, glutamate | During surgery and 8 weeks postoperative
  Analysis from muscle biopsies harvested from the vastus lateralis (muscle)
Pain receptors; glutamate receptors | During surgery and 8 weeks postoperative
  Analysis from muscle biopsies harvested from the vastus lateralis (muscle)

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Orthopaedic department, Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnsen M, Havik S, Husby VS, Winther SB, Foss OA, Husby OS, Lian OB. The use of tourniquet in total knee arthroplasty does not impact the functional outcome: a randomised controlled study. J Orthop Surg Res. 2024 Oct 30;19(1):704. doi: 10.1186/s13018-024-05203-y. PMID 39478609